CLINICAL TRIAL: NCT06720389
Title: Effect of Two Different Digital Construction Techniques of Implant-assisted Overdentures: a 3-year Prospective Radiographic Study
Brief Title: Effect of Two Different Digital Construction Techniques of Implant-assisted Overdentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A01010024RP
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Peri Implant Bone Loss
Keywords: Milled denture base; 3D-printing denture base,

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- milled mandibular overdenture opposed by maxillary complete denture (Active Comparator): A denture base milled from a pre-polymerized block of polymethylmethacrylate (Ivobase CAD) along with milled denture teeth from a block of tooth coloured material PMMA (SR Vivodent CAD).
  Interventions: Radiation: peri implant bone loss was assessed by CBCT; Other: posterior ridge resorption was assessed by CBCT
- 3D-Printed mandibular overdenture (Active Comparator): The printer (Rasdent 3d printer) was loaded with material of 3D-printed denture base and 3D- printed denture teeth (Dentca denture teeth shade A2). The mandibular denture teeth were printed as one unit then bonded to the lower printed denture base.
  Interventions: Radiation: peri implant bone loss was assessed by CBCT; Other: posterior ridge resorption was assessed by CBCT

INTERVENTIONS:
Radiation: peri implant bone loss was assessed by CBCT — using CBCT, vertical bone loss (VBL) was measured at baseline (T0), at1 year(T1), at 3 years(T3)
Other: posterior ridge resorption was assessed by CBCT — posterior ridge resorption was assessed by CBCT at baseline (T0), at 1 year( T1), at 3 years (T3). By superimposition of pre and post CBCT.

SUMMARY:
twenty patients received mandibular overdenture constructed by different construction techniques were classified equally and randomly into two groups peri implant bone loss was assessed by CBCT at baseline (T0), at1 year(T1), at 3 years(T3) and posterior ridge resorption was assessed by CBCT at baseline (T0), at 1 year( T1), at 3 years (T3). By superimposition of pre and post CBCT.

DETAILED DESCRIPTION:
twenty patients received mandibular overdenture constructed by different construction techniques were classified equally and randomly into two groups (n = 10 per group): Group A: received milled mandibular overdenture opposed by maxillary complete denture. Group B: received 3D-printed mandibular overdenture opposed by maxillary acrylic complete denture. peri implant bone loss was assessed by CBCT at baseline (T0), at1 year(T1), at 3 years(T3) and posterior ridge resorption was assessed by CBCT at baseline (T0), at 1 year( T1), at 3 years (T3). By superimposition of pre and post CBCT.

ELIGIBILITY:
Inclusion Criteria:

* All patient wearing maxillary conventional denture.
* All patients had temporary mandibular overdenture supported by vertically inserted 4-implant at least six months ago.
* A Cone Beam Computed Tomography (CBCT) done to verify the accurate position and success of the inserted implant.
* They were healthy, free from any systemic diseases relating to bone resorption such as uncontrolled diabetics or osteoporosis. This was achieved through medical history and clinical examination by physician.
* At least 15 mm restorative space must be available (from the mucosa covering the crest of the residual ridge to proposed occlusal plane) to permit construction of all types of tested prosthesis (class I according to Ahuja and Cagna). This was detected by a tentative jaw relation.
* All patients are of angel's class I maxillo-mandibular relationships.

Exclusion Criteria:

* Patients had head and neck radiotherapy, patients with bleeding disorders or hepatic patients.
* Patients with metabolic disorders as diabetes mellitus, osteoporosis and hepatic disorders that might affect osseointegration.
* Long term immunosuppress and corticosteroid drug therapy.
* Patient with abnormal habits as clenching and bruxism.
* Smoking patient.
* Uncooperative patients.
* Neuromuscular diseases.
* Patient with problems in TMJ.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-08-04 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
peri implant bone loss | at baseline (T0), at1 year(T1), at 3 years(T3)
  peri implant bone loss was assessed by CBCT
posterior ridge resorption | at baseline (T0), at 1 year( T1), at 3 years (T3).
  posterior ridge resorption was assessed by CBCT at baseline (T0), at 1 year( T1), at 3 years (T3). By superimposition of pre and post CBCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Khamisy NES, Emera RMK, Elmanci TM, Aboelez MA. Effect of two different digital construction techniques of mandibular implant-assisted overdentures on peri-implant bone loss and posterior ridge resorption: a 3-year prospective randomized clinical trial. BMC Oral Health. 2025 Jul 2;25(1):1040. doi: 10.1186/s12903-025-06425-0. PMID 40604700